CLINICAL TRIAL: NCT02001883
Title: Randomized Trial of the Association Between Low-Dose Statins and Nutraceuticals in High-intEnsity Statin-intoleRant patiENts With Very High Risk Coronary Artery diseasE
Brief Title: Low-dose Statins and Nutraceuticals in High-intensity Statin-intolerant Patients
Acronym: ADHERENCE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 807/2013/D-2
Record Dates: First submitted 2013-11-24; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease, nutraceuticals, statins
MeSH Terms: conditions — Coronary Artery Disease | interventions — Association; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Dietary Supplements; Simvastatin; Atorvastatin; policosanol; Berberine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Association low-dose statin and nutraceuticals (Active Comparator): Patients will receive the association between low-dose statin (10 to 20 mg/day of simvastatin or 5 to 10 mg/day atorvastatin) and a commercially available nutraceutical combined pill (1 capsule/day containing red yeast rice 200 mg, policosanol 10 mg, and berberine 500 mg).
  Interventions: Drug: Association low-dose statin and nutraceuticals
- Low-dose statin (Active Comparator): Patients will receive low-dose statin (10 to 20 mg/day of simvastatin or 5 to 10 mg/day atorvastatin)
  Interventions: Drug: Association low-dose statin and nutraceuticals

INTERVENTIONS:
Drug: Association low-dose statin and nutraceuticals
  Other Names: 10 to 20 mg/day of simvastatin; 5 to 10 mg/day atorvastatin; nutraceutical combined pill (1 capsule/day containing red yeast rice 200 mg, policosanol 10 mg, and berberine 500 mg).

SUMMARY:
The primary objective of this study is to compare the efficacy and tolerability of low-dose statin therapy vs. the association between a low-dose statin and a nutraceutical-based protocol in high-dose statin-intolerant patients with coronary artery disease deemed to be at high-risk.

DETAILED DESCRIPTION:
Several clinical trials have shown that in patients with atherosclerotic cardiovascular disease, reduction of low-density lipoprotein (LDL) level with a beta-hydroxy-beta-methylglutaryl coenzyme A reductase inhibitor (ie, statin) is associated with significant reductions in both mortality rate and major cardiac events.

Accordingly, current guidelines recommend that high-intensity statin therapy-such as rosuvastatin 20 to 40 mg or atorvastatin 80 mg-should be used to achieve at least a 50% reduction in LDL cholesterol unless otherwise contraindicated.

In real world clinical practice, however, high-intensity statin treatment is often discontinued by patients due to side effects. As alternatives, nonstatin drugs, such as ezetimibe, are often prescribed in association with moderate-to-low intensity statin.

It remains unknown, however, whether the association between moderate-to-low intensity statin therapy and and nutraceuticals (i.e. compounds derived from foods with cholesterol lowering actions) can have a therapeutic role in high-intensity statin-intolerant patients.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically-proven coronary artery disease
* Recent (<12 months) percutaneous coronary intervention
* Class I indication to receive statin treatment to achieve the LDL cholesterol goal of <70 mg/dL
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Long-term adherence to study treatments | Up to 12 months
  Satisfactory compliance (≥80%) in taking study drugs

SECONDARY OUTCOMES:
Number of participants with target LDL cholesterol | Up to 12 months
  Number of patients with at least a 50% reduction in LDL cholesterol as compared with baseline values at the end of the study period

CONTACTS AND LOCATIONS:
Locations (1):
- University Sapienza, Rome, Please Select, Italy